CLINICAL TRIAL: NCT06028958
Title: Effects Of Global Postural Re-Education And Neck Isometric Exercises In Patients With Cervical Radiculopathy
Brief Title: Global Postural Re-Education And Neck Isometric Exercises In Cervical Radiculopathy RADICULOPATHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-487-08-2023
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2023-08

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome accessor will be unaware of the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neck Isometrics Exercises (Active Comparator): This group of participants will receive neck isometric exercises along with routine physical therapy and a hot pack. In this regimen, the patient is commanded to apply minimal resistance on the physiotherapist's hand in front, back, and lateral positions. This resistance is applied for 10 sec with a 15 sec hold with 10-15 repetitions. The protocol will be given to the participants for two weeks. Each session will be of 40 minutes.
  Interventions: Other: Neck Isometrics Exercises
- Global Posture Re-Education (Experimental): This group of participants will receive the Global Posture Re-Education technique with a hot pack. The protocol will be given to the participants for two weeks (1 session on an alternative day with the home plan). Each session will be of 40 minutes.
  Interventions: Other: Global Posture Re-Education

INTERVENTIONS:
Other: Neck Isometrics Exercises — Isometric exercises are tightening (contractions) of a specific muscle or group of muscles. During isometric exercises, the muscle doesn't noticeably change length. The affected joint also doesn't move. Isometric exercises help maintain strength.
  Arms: Neck Isometrics Exercises
Other: Global Posture Re-Education — Global postural rehabilitation (GPR) is an approach that considers the body in its overall aspect. This technique aims to relax the envelope of the muscles (fascia) while relaxing the muscle chains to reduce the strain on the joints. The end result is a more suitable posture and less pain.
  Arms: Global Posture Re-Education

SUMMARY:
Cervical radiculopathy is a common neurological disorder that is caused by compression of the nerve, inflammation of nerve roots, or space-occupying lesions. Cervical radiculopathy is the most common health-related problem worldwide. The conservative approach like education, specific exercises, and spinal manipulation is usually given for chronic cases with good outcomes.

DETAILED DESCRIPTION:
Cervical Radiculopathy is a condition in which a nerve is entrapped between the bones and causes numbness and tingling. Neck isometric exercises are a basic treatment plan for strength training. Global postural reeducation is a technique the manual cervical traction along with body alignment that helps to reduce symptoms more rapidly. This whole procedure is completed more easily, without a machine and satisfying for the patient.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 35 years.
2. Both genders, Males and females
3. One-sided upper limb pain or numbness
4. Any 2 out of 4 tests are positive Spurling test, Distraction test, Ipsilateral cervical traction test, and Upper Limb test

Exclusion Criteria:

1. Bilateral upper limb pain
2. Previous history of cervical surgery
3. Cervical spine
4. Injection therapy in the past 2 weeks
5. Being Pregnant women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be measured at baseline, and change in pain intensity will be measured at 1st week, and 2nd week of treatment..
  Neck pain will be assessed utilizing the 10cm Visual Analogue Scale. The members will register their current pain level by selecting any from 0(no pain) to 10(unbearable pain) presented ahead a level line.
Level of Functional Disability | Change in Functional Status will be measured at baseline, at first week, and at second week of treatment.
  The level of Functional disability will be measured by using the neck disability index. It contains 10 readings including pain intensity, personal care, headache, lifting, reading, concentration, work, driving sleeping, and recreation. The questions are measured on a 6-point scale from 0 (no disability) to 5 (full disability). The numeric response for each item is summed for a score varying from 0 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Dr Ahmed, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: It will be shared soon after publication